CLINICAL TRIAL: NCT03228953
Title: Impact of Comprehensive Pharmacogenomic Testing on the Treatment of Major Depressive Disorder
Brief Title: Pharmacogenomic Testing in Major Depressive Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator retired.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AAAR4283
Record Dates: First submitted 2017-07-21; First posted 2017-07-25 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Major Depressive Disorder
Keywords: Pharmacogenomic testing; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacogenomic-guided therapy group (Experimental): In this group, results of pharmacogenomic testing will be provided to the treating physician within 2-5 working days. Thus, the patient's treatment provider will be able begin antidepressant adjustments based on pharmacogenomic testing report within a week of the baseline visit.
  Interventions: Other: Pharmacogenomic testing
- Treatment as usual (TAU) group (No Intervention): For patients randomized to this group, medication treatment decisions by the treating clinicians will be made without the availability of the pharmacogenomic report; however, the test results will be provided after the study completion to the patient treating physician.

INTERVENTIONS:
Other: Pharmacogenomic testing — Pharmacogenomic testing is delivered to treating providers of patients with major depressive disorder
  Arms: Pharmacogenomic-guided therapy group

SUMMARY:
This is a two-arm double-blind prospective randomized controlled trial (RCT) to evaluate clinical impact of pharmacogenomic testing on the treatment of major depressive disorder. Participants will be randomly assigned to two groups: pharmacogenomic-guided therapy group (guided group) and treatment as usual group (TAU group). The primary hypothesis is the pharmacogenomic-guided treatment group will demonstrate significantly higher percent improvement in depression score compared to treatment-as-usual group.

DETAILED DESCRIPTION:
To a large extent, variability in antidepressant efficacy can be explained by genetic variations that affect medication-metabolizing enzymes, drug transporters, and medication targets. Recent reviews demonstrated significant potential of pharmacogenomic testing in improving treatment of major depressive disorder. One of the major barriers towards successful implementation of pharmacogenomic testing for patients with major depressive disorder is lack of systematic evaluation of impact of this approach in routine clinical care settings. The major goal of this study is to systematically evaluate impact of comprehensive pharmacogenomic testing on the treatment of major depressive disorder in ambulatory setting.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of major depressive disorder (MDD)
2. Prescription of index antidepressant medications
3. Minimum score of 14 on the 17-item Hamilton Rating Scale for Depression (HAMD-17)

Exclusion Criteria:

1. Diagnosis of bipolar disorder (any type), schizophrenia, or schizoaffective disorders
2. Active diagnosis of substance abuse or dependence
3. Current suicidal ideation
4. Previous suicidal attempts
5. A person has already had pharmacogenetic testing done.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Score on the Hamilton Rating Scale for Depression (HAMD-17) | Up to 10 weeks
  The patient is rated by a clinician among 17 dimensions with a score on a 3 or 5 point scale. A score of 0-7 is considered to be normal. Scores of 20 or higher indicate moderate, severe, or very severe depression, and are usually required for entry into a clinical trial.

SECONDARY OUTCOMES:
Score on Subject-Rated 16-item Quick Inventory of Depression Symptomatology Scales (QIDS-SR) | Up to 10 weeks
  The Quick Inventory of Depressive Symptomatology is a short screening tool based on the larger Inventory of Depressive Symptomatology (IDS). Each item is scored on a scale from 0 to 3 points. Total scores range from 0 (no depression) to 27 (severe depression).
Score on the 9-item Patient Health Questionnaire (PHQ-9) | Up to 10 weeks
  The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Higher PHQ-9 scores are associated with decreased functional status and increased symptom-related difficulties, sick days and healthcare utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Cabrera, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No